CLINICAL TRIAL: NCT06096220
Title: Usage of 5-fluorouracil and Carnoy's Solution in Surgical Treatment of Odontogenic Keratocysts - Randomized, Controlled Clinical Study
Brief Title: Usage of 5-fluorouracil and Carnoy's Solution in Surgical Treatment of Odontogenic Keratocysts
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Miroslav Andric, Professor of Oral Surgery and Implantology, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36/17-2023
Record Dates: First submitted 2023-09-28; First posted 2023-10-23 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Odontogenic Keratocyst
MeSH Terms: conditions — Odontogenic Cysts | interventions — Eye Enucleation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Enucleation of OKC followed by local application of 5% 5-fluorouracil cream. Drug will be applied on the gauze left in the enucleation defect for 24 hours, after which the gauze will be removed.
  Interventions: Procedure: Enucleation; Diagnostic Test: incisional biopsy; Drug: Application of 5-fluorouracil
- Control group (Active Comparator): Enucleation of OKC followed by local application Carnoy solution. Carnoy solution will be applied into the cystic cavity for 5 minutes and bone defect will be treated by Carnoy solution for 3 minutes immediately after the enucleation.
  Interventions: Procedure: Enucleation; Diagnostic Test: incisional biopsy; Drug: Application of Carnoy solution

INTERVENTIONS:
Procedure: Enucleation — Enucleation is complete removal of the cyst from the bony defect of the jaw affected by the lesion. Osteotomy is performed to allow access to the cyst, cystic wall is detached from the bone and removed completely.
Diagnostic Test: incisional biopsy — Lesions clinically abd radiographically consistent with OKC will be submitted for histological examination to confirm the diagnosis of OKC
Drug: Application of 5-fluorouracil — 5% 5-fluorouracil cream will be applied immediately after the enucleation to the cystic cavity for 24 hours
  Arms: Experimental group
Drug: Application of Carnoy solution — Carnoy solution will be applied during the enucleation as described previously
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to compare surgical treatment outcomes of odontogenic keratocysts (OKC) treated with enucleation and local application of Carnoy's solution or 5% 5-fluorouracil. The main questions it aims to answer are:

1. What is the recurrence rate of OKC treated with enucleation and local application of 5% 5-fluorouracil cream in the period of three and five years after the treatment
2. What is the recurrence rate of OKC treated with enucleation and local application of Carnoy's solution in the period of three and five years after the treatment
3. Is there a difference in the recurrence rate between these two groups
4. What is the frequency of sensitivity disorders in the innervation zone of inferior alveolar and infraorbital nerves in both groups

Participants will be assigned to one of two groups after Histopathological verification (HP verification).They will be treated with enucleation and local application of Carnoy's solution or 5% 5-fluorouracil depending on group. After surgical treatment they will be monitored in accordance to standard treatment protocols for patients with OKC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified OKC of the upper or lower jaw;
* Indicated surgical treatment of OKC

Exclusion Criteria:

* Hypersensitivity to 5-fluorouracil and Carnoy's solution;
* Pathological fracture of the jaw in OKC region.
* Nevoid basal cell carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2028-06-10 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 5 years
  Number of participants with histologically verified OKC in site of previously treated OKC

SECONDARY OUTCOMES:
Sensitivity disorders | Immediately after the surgery up to one month
  dysesthesia and hypoesthesia in the surgical site

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Andric, Study Chair — University of Belgrade, School of Dental Medicine
Locations (1):
- School of Dental Medicine, Belgrade, Serbia